CLINICAL TRIAL: NCT04351789
Title: Impact of a Minimal Psychoeducational Intervention Versus Standard of Care on Anxiety Among Hospitalized COVID-19 Patients in Denmark: a Randomized Clinical Trial
Brief Title: Impact of a Minimal Psychoeducational Intervention on Anxiety Among Hospitalized COVID-19 Patients in Denmark
Acronym: PISCA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Responsible Party: Principal Investigator, Nina Weis, Professor, MD, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PISCA Study
Record Dates: First submitted 2020-04-11; First posted 2020-04-17 (Actual); Last update posted 2020-08-24 (Actual); Status verified 2020-08

CONDITIONS: COVID-19; Mental Health; Psychoeducation; Anxiety
MeSH Terms: conditions — COVID-19; Psychological Well-Being; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized 1:1 to either intervention group or control group
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the intervention, the RCT trial is not blinded, but the outcome measures are masked for health professionals and staff until the end of the study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Patients randomized to the intervention group will receive a minimal psychoeducational intervention just prior to discharge from the hospital. The goal of the intervention is that patients will be prepared and learn to interpret and react to physical and psychological symptoms that are related to recovering from a COVID-19 infection. The intervention is based on psychoeducational theory and consists of both written and verbal information. A manual describing the content and procedures of the intervention will be developed to ensure that the intervention is both replicable and transparent. The intervention has a planned duration of 30 minutes and will be conducted by a designated study affiliated researcher, who has a background in healthcare (i.e. nurse or medical doctor).
  Interventions: Other: Psychoeducational intervention
- Control Group (No Intervention): Standard of Care at discharge of patients with COVID-19 from hospital is to inform the patients whom to contact in case of worsening of the physical condition, such as increasing e.g. shortness of breath, and of precautions regarding further isolation to avoid infection of household and other contacts, if relevant. Information regarding the patient´s psychological condition is not part of a standard conversation at discharge.

INTERVENTIONS:
Other: Psychoeducational intervention — The written and verbal information provided at discharge to patients in the intervention arm will consist of:
  An explanation of the normal recovery period after hospitalization due to COVID-19. What can the patient expect physically, psychologically and emotionally, and what coping mechanism might be appropriate Social support in the recovery period and how this can be used constructively. In case of worsening of symptoms - physically or psychologically, where can the patient get help after discharge from hospital.
  These points are based on crisis psychology, enhancing the patients empowerment and self-management after discharge from hospital.
  Arms: Intervention Group

SUMMARY:
Background: There is limited knowledge on the psychological implications of COVID-19 among hospitalized patients and their close relatives. Moreover, evidence-based psychological interventions targeting hospitalized COVID-19 patients and their relatives are currently lacking.

Objective: To test a minimal psychoeducational intervention versus standard of care for reducing anxiety among hospitalized COVID-19 patients.

Methods and analysis: The trial is a Randomized Controlled Trial (RCT) with a 1 month and 3 month follow-up. Hospitalized COVID-19 patients are consecutively included at admission and randomized 1:1 to either an intervention or control group. Patients randomized to the intervention group will receive a minimal psychoeducational intervention just prior to discharge from the hospital. The goal of the intervention is that patients will be prepared and learn to interpret and react to physical and psychological symptoms that are related to recovering from a COVID-19 infection. Data is collected using standardized and validated patient reported outcome measures (PROMs) to assess mental health outcomes. The primary outcome is patient reported anxiety as assess by the Hospital Anxiety and Depression Scale.

Perspectives: This study will provide a comprehensive understanding of the psychological implications of the COVID-19 outbreak. If successful, the minimal intervention is easily implemented in daily clinical practice.

DETAILED DESCRIPTION:
INTRODUCTION Around 20% of people with COVID-19 becomes seriously ill with pneumonia and multi-organ failure, requiring hospital admission to relieve the symptoms and reduce mortality. To avoid any spreading of the virus, hospitalized COVID-19 patients are isolated. Thus, patients hospitalized with COVID-19 are limited in their social support and their only in-person contact is with healthcare staff in full personal protective equipment. Several studies highlight that isolation due to infection may have negative psychological implications. Moreover, Patients with confirmed or suspected COVID-19 may experience fear of the consequences of the infection. A high prevalence of persistent mental health problems has been found among patients during infectious disease outbreaks such as the 2003 outbreak of Severe Acute Respiratory Syndrome (SARS). Researchers and policy makers have highlighted that the psychological impact of the COVID-19 pandemic must be recognized alongside the physical symptoms for all those affected. Moreover, evidence-based evaluations and mental health interventions targeting hospitalized COVID-19 patients and their relatives are at present lacking. If left untreated, these psychological symptoms may have long-term health effects on patients and require treatment adding to the cost burden of managing the illness.

OBJECTIVE The objective of this project is to test the efficacy of a minimal psychoeducational intervention versus standard of care at discharge for reducing symptoms of anxiety in hospitalized patients during the COVID-19 outbreak

METHODS Design This is a Randomized Controlled Trial (RCT) among hospitalized COVID-19 patients.

Hypothesis The primary hypothesis is that a minimal psychological intervention will reduce anxiety as assessed by the Hospital Anxiety and Depression Scale (HADS) subscale for anxiety (HADS-A) by 1.5 points from baseline to follow-up 1 month after discharge from hospital. The estimated decrease in HADS-A is based on the clinically important difference found in patients with COPD and isolation studies.

Study population Patients will be recruited from the Department of Infectious Diseases and the COVID-19 isolation wards at Copenhagen University Hospital, Hvidovre; one of the major hospitals treating COVID-19 patients in Denmark.

Eligible patients are consecutively identified at time of admission. Included patients are randomized 1:1 to either a psychoeducational intervention or standard care delivered at discharge.

Sample size The primary outcome of interest is the intra-individual differences in HADS-A scores between baseline and follow-up 1 month post discharge. The design is paired with a power of 0.80 and an α at p=0.05. To identify a difference of 1.5 points, which is the minimal clinically important difference based on COPD and isolation studies, with an SD of 2.5 points, 25 patients are required in each group. Since the trial population consists of severely ill patients with high morbidity and mortality rates 2, approximately 30% of the sample are estimated to drop out. Thus, the RCT study requires 66 patients, with 33 in each group.

Intervention at discharge Patients randomized to the intervention group will receive a minimal psychoeducational intervention just prior to discharge from the hospital. The goal of the intervention is that patients will be prepared and learn to interpret and react to physical and psychological symptoms that are related to recovering from a COVID-19 infection. The intervention consists of both written and verbal information. While both the written and verbal information will be primarily targeted the patient, the role of relatives and their possible reactions will be part of the dialogue. A manual describing the content and procedures of the intervention will be developed to ensure that the intervention is both replicable and transparent. The intervention has a planned duration of 30 minutes and will be conducted by a designated study affiliated researcher, who has a background in healthcare (i.e. nurse or medical doctor).

Standard of care at discharge Standard of Care at discharge of patients with COVID-19 from hospital is to inform the patients whom to contact in case of worsening of the physical condition, such as increasing e.g. shortness of breath, and of precautions regarding further isolation to avoid infection of household and other contacts, if relevant. Information regarding the patient´s psychological condition is not part of a standard conversation at discharge.

Blinding Due to the nature of the intervention, the RCT trial is not blinded, but the outcome measures are masked for health professionals and staff until the end of the study.

Data collection Data is collected using standardized questionnaires at four timepoints; baseline completed within 48 hours after admission (T0), at discharge, but prior to intervention (T1), 1 month (T2), 3 months (T3), and 12 months (T4). Patients will answer the questionnaires electronically in REDCap© or via phone interview conducted by a study nurse or medical student. Clinical data is collected from the medical records and entered into the REDCap© database.

The following internationally well validated PROMs will be used to assess mental health/distress:

* Anxiety and depression will be assessed using the Danish version of the HADS. The primary outcome in the RCT study is anxiety measured by HADS-A.
* Perceived stress is measured using the Perceived Stress Scale - 10 item (PSS-10).
* Harvard Trauma Questionnaire (HTQ) is used to assess subjective distress caused by traumatic events.
* Health related quality of life is measured by SF-12, a short version of the Medical Outcomes Study (MOS) 36-item Short-Form Health Survey SF-36.

Sociodemographic and clinical variables The following demographic and clinical data are collected from the patients records: age, gender, marital status, residence in nursing home, medicine, smoking status, BMI, previous history of psychiatric illness, physical symptoms, and clinical parameters such as Temperature (>/> 38C); demand of oxygen support (< 5 litres O2/minute; 5-10 litres O2/minute; >10-30 O2/minute or need for mechanical ventilation). Biochemical parameters (Hemoglobin, White Blood Cell (WBC) count, lymphocyte count, Lactate Dehydrogenase, Alanine Amino Transferase (ALT), CRP). Length of hospital stay is collected at discharge. Information regarding contact to general practitioner and current psychological treatment outside of the study is collected during follow-up.

Statistical analysis Descriptive statistics of demographic characteristics at baseline (T0) will be computed. The primary analysis for the RCT study will be performed on the basis of the intention-to-treat principle. Baseline data for the two groups will be compared with Student's t test, the chi-square test, or nonparametric tests. To analyse within group differences in outcome scores, a Student´s t test or Wilcoxon rank-sum test will be used. A mixed regression model will be used to assess the change within-group and between groups over time. The co-variables included in the models will be chosen based on an a priori hypothesis, the bivariate analysis and clinical relevance. Analyses will be performed using the STATA 13 software and in collaboration with an experienced statistician. All reported p-values are two-sided using a significance level of 0.05.

ETHICAL CONSIDERATIONS The study has been approved by the Danish Data Protection Agency [P-2020-349]. The national Health Research Ethics Committee has assessed the intervention as not being a significant biomedical intervention [jr. nr. 20025879]. All participating patients will provide written informed consent before any data collection.

TIME SCHEDULE This is a two-year study initiated as soon as possible and no later than mid April 2020.

DISSIMINATION Publication of positive, neutral or negative results in international, peer-reviewed journals will be sought. In addition, results will be communicated at relevant scientific meetings and conferences.

PERSPECTIVE The results from this study have a number of important potential implications. First, by quantifying the magnitude of psychiatric symptoms among hospitalized COVID-19 patients, potential risk factors associated with these symptoms can be identified. Second, there is a need to develop and test the efficacy of minimal psychological intervention for reducing psychiatric morbidity among COVID-19 patients. Providing psychological treatment and support may reduce the burden of comorbid mental health conditions both short and long-term. The challenge is to provide mental health services in the context of patient isolation. Hence, the intervention is designed to give healthcare professionals an instrument that is clinically applicable and easy to implement even in isolated patients. Finally, the longitudinal design of the study capturing experiences over time, can be used to identify when in the trajectory psychological interventions are most needed.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years of age
* In-hospitalized with confirmed COVID-19 diagnosis,
* HADS-A score ≥8
* Able to read and understand Danish,
* Able to provide written informed consent

Exclusion Criteria:

* Patients with pulmonary cancer
* Patients who are terminally ill

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
Anxiety 1 month | 1 month post discharge
  Anxiety measured by the Hospital Anxiety and Depression Scale. Range in score: 0 - 28. Higher scores = more symptoms of anxiety.

SECONDARY OUTCOMES:
Anxiety 3 months | 3 months post discharge
  Anxiety measured by the Hospital Anxiety and Depression Scale. Range in score: 0 - 28. Higher scores = more symptoms of anxiety.
Depression 3 months | 3 months post discharge
  Depression measured by the Hospital Anxiety and Depression Scale. Range in score: 0 - 28. Higher scores = more symptoms of depression.
Post Traumatic Stress Disorder (PTSD) symptoms 3 months | 3 months post discharge
  PTSD symptoms measured by the Harvard Trauma Questionnaire. Range in score: 16 - 64. Higher scores = more symptoms of PTSD
Anxiety 12 months | 12 months post discharge
  Anxiety measured by the Hospital Anxiety and Depression Scale. Range in score: 0 - 28. Higher scores = more symptoms of anxiety.
Post Traumatic Stress Disorder (PTSD) symptoms 12 months | 12 months post discharge
  PTSD symptoms measured by the Harvard Trauma Questionnaire. Range in score: 16 - 64. Higher scores = more symptoms of PTSD
Depression 12 months | 12 months post discharge
  Depression measured by the Hospital Anxiety and Depression Scale. Range in score: 0 - 28. Higher scores = more symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Weis, MD, PhD, Principal Investigator — Copenhagen University Hospital, Hvidovre
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researchers due to regulatory restrictions.

REFERENCES:
- [Background] Weiss P, Murdoch DR. Clinical course and mortality risk of severe COVID-19. Lancet. 2020 Mar 28;395(10229):1014-1015. doi: 10.1016/S0140-6736(20)30633-4. Epub 2020 Mar 17. No abstract available. PMID 32197108
- [Background] Purssell E, Gould D, Chudleigh J. Impact of isolation on hospitalised patients who are infectious: systematic review with meta-analysis. BMJ Open. 2020 Feb 18;10(2):e030371. doi: 10.1136/bmjopen-2019-030371. PMID 32075820
- [Background] Dashiell-Earp CN, Bell DS, Ang AO, Uslan DZ. Do physicians spend less time with patients in contact isolation?: a time-motion study of internal medicine interns. JAMA Intern Med. 2014 May;174(5):814-5. doi: 10.1001/jamainternmed.2014.537. No abstract available. PMID 24686899
- [Background] Sharma A, Pillai DR, Lu M, Doolan C, Leal J, Kim J, Hollis A. Impact of isolation precautions on quality of life: a meta-analysis. J Hosp Infect. 2020 May;105(1):35-42. doi: 10.1016/j.jhin.2020.02.004. Epub 2020 Feb 12. PMID 32059996
- [Background] Xiang YT, Yang Y, Li W, Zhang L, Zhang Q, Cheung T, Ng CH. Timely mental health care for the 2019 novel coronavirus outbreak is urgently needed. Lancet Psychiatry. 2020 Mar;7(3):228-229. doi: 10.1016/S2215-0366(20)30046-8. Epub 2020 Feb 4. No abstract available. PMID 32032543
- [Background] Maunder R, Hunter J, Vincent L, Bennett J, Peladeau N, Leszcz M, Sadavoy J, Verhaeghe LM, Steinberg R, Mazzulli T. The immediate psychological and occupational impact of the 2003 SARS outbreak in a teaching hospital. CMAJ. 2003 May 13;168(10):1245-51. PMID 12743065
- [Background] Lam MH, Wing YK, Yu MW, Leung CM, Ma RC, Kong AP, So WY, Fong SY, Lam SP. Mental morbidities and chronic fatigue in severe acute respiratory syndrome survivors: long-term follow-up. Arch Intern Med. 2009 Dec 14;169(22):2142-7. doi: 10.1001/archinternmed.2009.384. PMID 20008700
- [Background] Lee AM, Wong JG, McAlonan GM, Cheung V, Cheung C, Sham PC, Chu CM, Wong PC, Tsang KW, Chua SE. Stress and psychological distress among SARS survivors 1 year after the outbreak. Can J Psychiatry. 2007 Apr;52(4):233-40. doi: 10.1177/070674370705200405. PMID 17500304
- [Background] Kwek SK, Chew WM, Ong KC, Ng AW, Lee LS, Kaw G, Leow MK. Quality of life and psychological status in survivors of severe acute respiratory syndrome at 3 months postdischarge. J Psychosom Res. 2006 May;60(5):513-9. doi: 10.1016/j.jpsychores.2005.08.020. PMID 16650592
- [Background] Mak IW, Chu CM, Pan PC, Yiu MG, Ho SC, Chan VL. Risk factors for chronic post-traumatic stress disorder (PTSD) in SARS survivors. Gen Hosp Psychiatry. 2010 Nov-Dec;32(6):590-8. doi: 10.1016/j.genhosppsych.2010.07.007. Epub 2010 Sep 15. PMID 21112450
- [Background] Shigemura J, Ursano RJ, Morganstein JC, Kurosawa M, Benedek DM. Public responses to the novel 2019 coronavirus (2019-nCoV) in Japan: Mental health consequences and target populations. Psychiatry Clin Neurosci. 2020 Apr;74(4):281-282. doi: 10.1111/pcn.12988. Epub 2020 Feb 23. No abstract available. PMID 32034840
- [Background] Zandifar A, Badrfam R. Iranian mental health during the COVID-19 epidemic. Asian J Psychiatr. 2020 Jun;51:101990. doi: 10.1016/j.ajp.2020.101990. Epub 2020 Mar 4. No abstract available. PMID 32163908
- [Background] Zhou X, Snoswell CL, Harding LE, Bambling M, Edirippulige S, Bai X, Smith AC. The Role of Telehealth in Reducing the Mental Health Burden from COVID-19. Telemed J E Health. 2020 Apr;26(4):377-379. doi: 10.1089/tmj.2020.0068. Epub 2020 Mar 23. No abstract available. PMID 32202977
- [Background] Puhan MA, Frey M, Buchi S, Schunemann HJ. The minimal important difference of the hospital anxiety and depression scale in patients with chronic obstructive pulmonary disease. Health Qual Life Outcomes. 2008 Jul 2;6:46. doi: 10.1186/1477-7525-6-46. PMID 18597689
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Bjelland I, Dahl AA, Haug TT, Neckelmann D. The validity of the Hospital Anxiety and Depression Scale. An updated literature review. J Psychosom Res. 2002 Feb;52(2):69-77. doi: 10.1016/s0022-3999(01)00296-3. PMID 11832252
- [Background] Herrmann C. International experiences with the Hospital Anxiety and Depression Scale--a review of validation data and clinical results. J Psychosom Res. 1997 Jan;42(1):17-41. doi: 10.1016/s0022-3999(96)00216-4. PMID 9055211
- [Background] Butler AC, Chapman JE, Forman EM, Beck AT. The empirical status of cognitive-behavioral therapy: a review of meta-analyses. Clin Psychol Rev. 2006 Jan;26(1):17-31. doi: 10.1016/j.cpr.2005.07.003. Epub 2005 Sep 30. PMID 16199119
- [Background] Schnyder U, Ehlers A, Elbert T, Foa EB, Gersons BP, Resick PA, Shapiro F, Cloitre M. Psychotherapies for PTSD: what do they have in common? Eur J Psychotraumatol. 2015 Aug 14;6:28186. doi: 10.3402/ejpt.v6.28186. eCollection 2015. PMID 26290178
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Eskildsen A, Dalgaard VL, Nielsen KJ, Andersen JH, Zachariae R, Olsen LR, Jorgensen A, Christiansen DH. Cross-cultural adaptation and validation of the Danish consensus version of the 10-item Perceived Stress Scale. Scand J Work Environ Health. 2015 Sep 1;41(5):486-90. doi: 10.5271/sjweh.3510. Epub 2015 Jun 25. PMID 26111225
- [Background] Mollica RF, Caspi-Yavin Y, Bollini P, Truong T, Tor S, Lavelle J. The Harvard Trauma Questionnaire. Validating a cross-cultural instrument for measuring torture, trauma, and posttraumatic stress disorder in Indochinese refugees. J Nerv Ment Dis. 1992 Feb;180(2):111-6. PMID 1737972
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Bjorner JB, Thunedborg K, Kristensen TS, Modvig J, Bech P. The Danish SF-36 Health Survey: translation and preliminary validity studies. J Clin Epidemiol. 1998 Nov;51(11):991-9. doi: 10.1016/s0895-4356(98)00091-2. PMID 9817117
- See also: World Health Organisation. Q&A on coronaviruses (COVID-19) — http://www.who.int/news-room/q-a-detail/q-a-coronaviruses